## Clinical Performance of Two Reusable Silicone Hydrogel Contact Lenses

STUDY ID CLL949-C024

**PROTOCOL** 

NCT05766787



#### **Device Protocol for CLL949-C024**

Title: Clinical Performance of Two Reusable Silicone Hydrogel Contact

Lenses

Protocol Number: CLL949-C024

Clinical Investigation

Interventional

Type:

Test Product: Alcon serafilcon A contact lenses

Sponsor Name and Alcon Research, LLC, and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Property of Alcon Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Alcon

Document ID: V-CLN-0035929


Status: Approved, Version: 3.0 Approved Date: 13 Apr 2023

#### Investigator Agreement:

- I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices; applicable international and national regulations, laws, guidelines, and standards; the conditions of approval imposed by the reviewing IRB or regulatory authority; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current investigator's brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authority? | | |
|---|---|---|---|
| | □ No | □Yes | |
| | Have you | ever been involved in a study or other r | esearch that was terminated? |
| | □ No | □Yes | |
| | If yes, ple | ease explain here: | |
| Pr | incipal inve | estigator: | |
| | | Signature | Date |
| | ame and prosition: | ofessional | |
| A | ldress: | | |

#### **Table of Contents**

| De | vice Prote | ocol for CLL949-C024 | 1 |
|---|---|---|---|
| Ta | ble of Co | ntents | 3 |
| Lis | st of Table | es | 5 |
| Lis | st of Figu | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OF | F ACRONYMS AND ABBREVIATIONS | 13 |
| 3 | PROTO | COL SUMMARY | 15 |
| 4 | PROTO | COL AMENDMENTS | 29 |
| 5 | INTROI | DUCTION | 29 |
| | 5.1 | Rationale and Background | 29 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | |
| 6 | STUDY | OBJECTIVES | 31 |
| | 6.1 | Primary Objective(s) | 31 |
| | 6.2 | Secondary Objective(s) | 31 |
| | 6.4 | Safety Objective(s) | |
| 7 | INVES 7 | TIGATIONAL PLAN | 35 |
| | 7.1 | Study Design | 35 |
| | 7.2 | Rationale for Study Design | 35 |
| | | 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations | 37 |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | |
| | 7.4 | Rationale for Choice of Comparator Product | 37 |
| | 7.5 | Data Monitoring Committee | 37 |
| 8 | STUDY | POPULATION | 37 |
| | 8.1 | Inclusion Criteria | 38 |
| | 8.2 | Exclusion Criteria | 39 |
| | 8.3 | Rescreening of Subjects | |
| 9 | TREAT | MENTS ADMINISTERED | 40 |

| | 9.1 | Investigational Product(s) | 40 |
|---|---|---|---|
| | 9.2 | Other Medical Device or Medication Specified for Use During the Study | 44 |
| | 9.3 | Treatment Assignment / Randomization | 44 |
| | 9.4 | Treatment masking | 45 |
| | 9.5 | Accountability Procedures | 46 |
| | 9.6 | Changes to concomitant medications, treatments/ procedures | 47 |
| 10 | STUDY | PROCEDURES AND ASSESSMENTS | 47 |
| | 10.1 | Informed Consent and Screening | 48 |
| | 10.2 | Description of Study Procedures and Assessments | 49 |
| | | 10.2.1 Demographics | |
| | | 10.2.2 Medical History | |
| | | 10.2.3 Investigational Product Compliance | 49 |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 49 |
| | | 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment | 49 |
| | | 10.2.6 Device Deficiencies: Safety Assessment | 50 |
| | | 10.2.7 Best Corrected Visual Acuity: Safety Assessment | |
| | | 10.2.8 Additional Study Assessments | |
| | 10.3 | Unscheduled Visits | 50 |
| | 10.4 | Discontinued Subjects | 51 |
| | | 10.4.1 Screen Failures | 51 |
| | | 10.4.2 Discontinuations | 51 |
| | | 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product | 51 |
| | 10.5 | Clinical Study Termination | 52 |
| | | 10.5.1 Follow-Up of Subjects After Study Participation has Ended | 52 |
| 11 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 52 |
| | 11.1 | General Information | 52 |
| | 11.2 | Monitoring for Adverse Events | 55 |
| | 11.3 | Procedures for Recording and Reporting | 56 |
| | 11.4 | Return Product Analysis | 58 |
| | 11.5 | Unmasking of the Study Treatment | 58 |
| | 11.6 | Follow-Up of Subjects with Adverse Events | |
| | 11.7 | Pregnancy in the Clinical Study | |
| 12 | | SIS PLAN | 59 |

| 12.1 | Subject Evaluability | |
|-----------|------------------------------------------------------|----|
| 12.2 | Analysis Sets. | 59 |
| | 12.2.1 Safety Analysis Set | 59 |
| | 12.2.2 Full Analysis Set | 60 |
| | 12.2.3 Per Protocol Analysis Set | |
| 12.3 | Demographic and Baseline Characteristics | 60 |
| 12.4 | Effectiveness Analyses | 60 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 60 |
| | 12.4.1.1 Statistical Hypotheses | |
| | 12.4.1.2 Analysis Methods | 61 |
| 12.5 | Handling of Missing Data | 65 |
| 12.6 | Safety Analyses | 65 |
| 12.7 | Interim Analyses and Reporting | 66 |
| 12.8 | Sample Size Justification. | 66 |
| 13 DATA H | ANDLING AND ADMINISTRATIVE REQUIREMENTS | 68 |
| 13.1 | Subject Confidentiality | 68 |
| 13.2 | Completion of Source Documents and Case Report Forms | 68 |
| 13.3 | Data Review and Clarifications | 69 |
| 13.4 | Sponsor and Monitoring Responsibilities | 69 |
| 13.5 | Regulatory Documentation and Records Retention | 70 |
| 13.6 | Quality Assurance and Quality Control | 70 |
| 14 ETHICS | | |
| 15 REFERE | NCES | 72 |
| 15.1 | Regulations and Standards | 72 |
| 13.1 | regulations and Standards | /2 |

 Figure 11-1

Figure 11-2

Categorization of All Adverse Events......53

#### 1 GLOSSARY OF TERMS

| Names of Test Product(s) | Throughout this document, test product(s) will be referred to as Alcon serafilcon A contact lenses |
|---|---|
| Name of Comparator<br>Product(s) | ACUVUE® OASYS with HYDRACLEAR® PLUS Technology |
| Adverse Device Effect (ADE) | Adverse event related to the use of an investigational medical device or comparator. |
| | Note: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation; any malfunction; and use error or intentional misuse. |
| Adverse Event (AE) | Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device or comparator and whether anticipated or unanticipated. |
| | Note: For subjects, this definition includes events related to the investigational medical device, comparator, or the procedures involved. For users or other persons, this definition is restricted to the use of the investigational medical device or comparator. |
| | Requirements for reporting Adverse Events in the study can be found in Section 11. |
| Anticipated Serious Adverse Device Effect (ASADE) | An effect which by its nature, incidence, severity, or outcome has been identified in the risk assessment. |

| Clinical Investigation Plan (CIP) | The document(s) stating the rationale, objectives, design, and prespecified analysis, methodology, organization, monitoring, conduct, and record-keeping of the clinical investigation. Note: The protocol and other documents referenced in the protocol (for example, the Statistical Analysis Plan, the Manual of Procedures, the Deviations and Evaluability Plan, and the Protocol Monitoring Plan) comprise the CIP. |
|---|---|
| Clinical Investigation | The document describing the design, execution, statistical |
| Report (CIR) / Clinical | analysis, and results of a clinical investigation. The Clinical |
| Study Report | Investigation Report is synonymous with the Clinical Study Report. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance. |
| | Note: This definition includes malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling related to the investigational medical device or the comparator. |
| | Requirements for reporting Device Deficiencies in the study can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for participation in the study. |
| Point of Enrollment | The time at which, following recruitment and before any |
| | clinical investigation-related procedures are undertaken, a subject signs and dates the informed consent form. |

| Interventional Clinical Trial | A pre- or postmarket clinical investigation where the |
|---|---|
| | assignment of a subject to a particular medical device is |
| | decided in advance by a clinical investigation plan, or |
| | diagnostic or monitoring procedures requested in the CIP are |
| | in addition to those available as normal clinical practice and |
| | burden the subject. |
| Investigational Product | A preventative (vaccine), a therapeutic (drug or biologic), |
| | device, diagnostic, or palliative used as a test or comparator |
| | product in a clinical trial, including a product with a |
| | marketing authorization when used or assembled |
| | (formulated or packaged) in a way different from the |
| | authorized form, or when used for an unauthorized |
| | indication, or when used to gain further information about |
| | the authorized form. |
| Malfunction | Failure of an investigational medical device to perform in |
| | accordance with its intended purpose when used in |
| | accordance with the instructions for use or clinical |
| | investigation plan (CIP), or investigator's brochure (IB). |
| Nonserious Adverse Event | Adverse event that does not meet the criteria for a serious |
| | adverse event. |
| 7 1 1 1 1 1 1 1 | |
| Randomized Subject | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |
| Elicu (SADE) | consequences characteristic of a serious adverse event. |
| | 1 |

## Serious Adverse Event (SAE)

Adverse event that led to any of the following:

- Death.
- A serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
  - a) a life-threatening illness or injury

    Note: Life-threatening means that the individual was
    at immediate risk of death from the event as it
    occurred, i.e., it does not include an event which
    hypothetically might have caused death had it
    occurred in a more severe form.
  - b) any potentially sight-threatening event or permanent impairment to a body structure or a body function including chronic diseases.
  - c) inpatient hospitalization or prolonged hospitalization.
  - d) a medical or surgical intervention to prevent a) or b).
  - e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.
- Fetal distress, fetal death, congenital abnormality or birth defect including physical or mental impairment.

Note: Planned hospitalization for a preexisting condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event.

Refer to Section 11 for additional SAEs.

| Serious Health Threat | Signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users, or other persons, and that requires prompt remedial action for other subjects, users, or |
|---|---|
| | Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals. |
| Significant Nonserious Adverse Event | A significant non-serious adverse event is a symptomatic, device-related, non-sight-threatening adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 11 for additional Significant Nonserious AEs. |
| Study Start | The start of the study is considered to coincide with the enrollment of the first patient. |
| Study Completion | The completion of the study is considered to coincide with the study-level last subject last visit or the decision to terminate the trial, whichever is later. |
| Unanticipated Serious Adverse Device Effect (USADE) | Serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the risk assessment. |

| Use Error | User action or lack of user action while using the medical |
|---|---|
| | device that leads to a different result than that intended by |
| | the manufacturer or expected by the user. |
| | Note: |
| | a) Use error includes the inability of the user to complete a task. |
| | b) Use errors can result from a mismatch between the characteristics of the user, user interface, task, or use environment. |
| | c) Users might be aware or unaware that a use error has occurred. |
| | d) An unexpected physiological response of the patient |
| | is not by itself considered a use error. |
| | e) A malfunction of a medical device that causes an |
| | unexpected result is not considered a use error." |

#### 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2–1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| ADE | Adverse device effect |
| AE | Adverse event |
| AOHP | ACUVUE® OASYS with HYDRACLEAR® PLUS Technology |
| ASADE | Anticipated serious adverse device effect |
| BCVA | Best corrected visual acuity |
| CFR | Code of Federal Regulations |
| CIP | Clinical investigation plan |
| CIR | Clinical investigation report |
| COL | Clinical Operations Lead |
| CRF | Case report form |
| CSM | Clinical Site Manager |
| CTT | Clinical Trial Team |
| D | Diopter |
| DEP | Deviations and evaluability plan |
| Diff | difference |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| EN | European Standard |
| FAS | Full analysis set |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| LogMAR | Logarithm of the minimum angle of resolution |
| mm | millimeter |
| MOP | Manual of procedures |
| N | Number of subjects |
| N/A | Not applicable |
| NI | Noninferiority |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |
| PP | Per Protocol |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |

Document ID: V-CLN-0035929

| Abbreviation | Definition |
|--------------|---------------------------------------------|
| SD | Standard deviation |
| Seq | sequence |
| SLE | Slit lamp examination |
| SOP | Standard operating procedure |
| UCL | Upper confidence limit |
| US | United States |
| USADE | Unanticipated serious adverse device effect |
| VA | Visual acuity |

#### **3 PROTOCOL SUMMARY**

| Investigational | Device |
|---|---|
| product type | |
| Study type | Interventional |
| Investigational | Test Product: Alcon serafilcon A contact lenses (LID022821) |
| products | Comparator Product: ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses |
| Purpose and | The purpose of this study is to assess the clinical performance of the |
| Scientific | investigational Alcon serafilcon A contact lenses as compared to |
| Rationale for | marketed ACUVUE® OASYS with HYDRACLEAR® PLUS |
| the Study | Technology contact lenses when worn on a daily wear modality. |
| | The design of this study is |
| | justified based upon preclinical and clinical testing, as described within |
| | the investigator's brochure. AOHP contact lenses were chosen as the |
| | comparator product because these lenses also are reusable contact lenses |
| | (see Package Insert for AOHP contact lenses). Subjects will be provided |
| | with CLEARCARE® Cleaning & Disinfecting Solution to use with the |
| | study lenses. |

| Brief | This study aims to compare the clinical performance |
|---|---|
| Summary of | at the end of the |
| the Protocol | replacement cycles of Alcon serafilcon A contact lenses compared to ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses, when worn on a daily wear modality. Volunteer subjects aged 18 or over who are habitual spherical soft contact lens wearers (excluding current/previous AOHP habitual lens wearers and daily disposable lens wearers), have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 8 hours per day, will be included. This is a prospective, randomized, double-masked, bilateral, crossover study. The expected outcome of this study is to demonstrate noninferiority in the visual acuity at distance when wearing Alcon serafilcon A contact lenses compared to AOHP contact lenses |
| Objective(s) | The primary objective of this study is to demonstrate noninferiority in the visual acuity at distance when wearing Alcon serafilcon A contact lenses compared to ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses when worn on a daily wear modality. |
| | The safety objective is to describe the safety profile of the study products. |
| Endpoint(s) | Primary Efficacy |
| | Distance visual acuity (logMAR) with study lenses at Week 1 |





# Safety Adverse events Biomicroscopy findings Device deficiencies Assessment(s) Effectiveness BCVA (logMAR distance with manifest refraction) Manifest refraction Distance visual acuity (logMAR) with study lenses Safety Adverse events Biomicroscopy Device deficiencies

| Study Design | This will be a multisite, prospective, randomized, double masked, bilateral, crossover study comparing 2 reusable soft contact lenses. The expected duration of subject participation in the study is approximately 28 days (~14 days per each lens type), with 7 scheduled visits. Subjects will be asked to wear their habitual spectacles only (no contact lens wear) during the washout periods for 2 (at least 48 hours) to 4 days after Visit 1 and after Visit 4. |
|---|---|
| Subject<br>population | Planned number of subjects enrolled/consented: ~185 Planned number of completed subjects: 168 |
| Sites and<br>Locations | Planned number of clinical sites: ~ 14 Planned locations (initial list of locations, which may change during start up or conduct according to study needs): US |
| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.</li> <li>Manifest cylinder of ≤ -0.75 D in each eye.</li> <li>Best corrected visual acuity (BCVA) 20/25 Snellen (0.10 logMAR) or better in each eye.</li> </ul> |
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) | <ul> <li>Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.</li> <li>Habitual AOHP contact lens wearers and current habitual wearers of any daily disposable contact lenses.</li> </ul> |
| Data analysis<br>and sample<br>size<br>justification | Planned Data Analysis |

| | Endpoint | Comparison | Statistical Model |
|---|---|---|---|
| | Primary | Comparison | Statistical Model |
| | Distance VA | Alcon serafilcon A<br>contact lenses vs<br>AOHP contact<br>lenses | Mixed effects repeated measures NI margin = 0.05 (logMAR) |
| | 0 10 1 | | |
| | Sample Size J | | |
| | | lculation is based on a | |
| | which evaluate | d performance of Alco | on serafilcon A contact lenses and |
| | AOHP contact | lenses. | |
| 1 | | | |

# Associated materials

- CLEARCARE® Cleaning & Disinfecting Solution supplied by sponsor to be provided to subjects for use during the study.
- Lubrication/rewetting drops will not be permitted.
- CLEARCARE® Plus with Hydraglyde Cleaning & Disinfecting Solution is not recommended.

Table 3-1 Schedule of Study Procedures and Assessment

| | | | Lens 1<br>(Period 1) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after Visit 1)] | Visit 3<br>Week 1<br>Follow-up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 2] | Visit 4<br>Week 2<br>Follow- up<br>Lens 1<br>[7-0/+ 1<br>days after<br>Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4)] | Visit 6<br>Week 1<br>Follow-up<br>Lens 2<br>[7-0/+ 1<br>days after<br>Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| Informed Consent | | X | | | | | | | | |
| Demographics | | X | | | | | | | | |
| Medical History | | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medications | | X | X | X | X | X | X | X | X | X |
| Inclusion/ Exclusion | | X | | | | | | | | |
| Habitual lens<br>(brand, lens<br>power, lens<br>care) | | X | | | | | | | | |
| In office subjective questionnaire Habitual lens wear and rewetting drop usage | | Х | | | | | | | | |
| Keratometry | | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |

| | | | Lens 1<br>(Period 1) | | | Lens 2<br>(Period 2) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after Visit 1)] | Visit 3<br>Week 1<br>Follow-up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 2] | Visit 4 Week 2 Follow- up Lens 1 [7 -0/+ 1 days after Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4)] | Visit 6 Week 1 Follow-up Lens 2 [7 -0/+ 1 days after Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| VA w/ habitual<br>correction <sup>+</sup><br>(OD, OS,<br>logMAR<br>distance)* | | Х | | | | | | X | X | (X) |
| Manifest refraction* | | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| BCVA (OD, OS,<br>logMAR distance with<br>manifest refraction) | | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| Biomicroscopy | | X | X | X | X | X | X | X | X | X |

| | | | Len<br>(Peri | od 1) | | | Lens 2<br>(Period 2) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after Visit 1)] | Visit 3<br>Week 1<br>Follow-up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 2] | Visit 4 Week 2 Follow- up Lens 1 [7 -0/+ 1 days after Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4)] | Visit 6 Week 1 Follow-up Lens 2 [7 -0/+ 1 days after Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| Fitting of investigational products (trial assessments): (Test and Comparator)* - VA (logMAR distance) - Lens movement (Overall fit- primary and peripheral gazes) - Lens position (Centration) | | X | | | | | | | | |
| Randomization | | X | | | | | | | | |
| Dispense study lenses | | | X | X | | X | X<br>X | | | (X) |
| VA w/study lenses,<br>(OD, OS, logMAR | | | X | X | X | X | X | X | (X) | (X) |

| | | | Lens 1<br>(Period 1) | | | Lens 2<br>(Period 2) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after | Visit 3 Week 1 Follow-up Lens 1 [7 -0/+ 1 days after Visit 2] | Visit 4 Week 2 Follow- up Lens 1 [7 -0/+ 1 days after Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after | Visit 6 Week 1 Follow-up Lens 2 [7 -0/+ 1 days after Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |

| | | | Ler<br>(Peri | od 1) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after | Visit 3<br>Week 1<br>Follow-up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 2] | Visit 4<br>Week 2<br>Follow- up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after | Visit 6<br>Week 1<br>Follow-up<br>Lens 2<br>[7 -0/+ 1<br>days after<br>Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| AEs α | | X | X | X | X | X | X | X | X | X |
| Device deficiencies | | X | X | X | X | X | X | X | X | X |
| Exit Form | | (X) | (X) | (X) | (X) | (X) | (X) | X | X | (X) |

Document ID: V-CLN-0035929 Status: Approved, Version: 3.0 Approved Date: 13 Apr 2023 

| (X) Assessment performed as necessary, e.g., decrease of VA by 2 lines or more with investigational product (IP) |
|---|
| Source only (source transferred to the sponsor upon request) |
| a Comprehensive details of all AEs will be documented in the source records, however limited collection will be utilized in the eCRF (see MOP for details |

#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the study sponsor and must be approved by the IRB/IEC and global and regional health authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

Refer to Appendix A for detailed description of amendments.

#### 5 INTRODUCTION

#### 5.1 Rationale and Background

The investigational contact lens (Alcon serafilcon A) is intended for the optical correction of refractive ametropia in persons with nondiseased eyes. This study will evaluate the on-eye clinical performance of investigational Alcon serafilcon A contact lenses compared against marketed ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses to evaluate product performance in the intended population, when worn on a daily wear modality.

ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses were chosen as the comparator product because these lenses also are reusable contact lenses (see Package Insert for ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses). The intended use of this contact lens is vision correction; therefore, the measurement of distance VA is planned as the primary effectiveness endpoint.

#### 5.2 Purpose of the Study

The purpose of this study is to assess the clinical performance of the investigational Alcon serafilcon A contact lenses as compared to marketed ACUVUE® OASYS with HYDRACLEAR® PLUS Technology contact lenses. The primary objective of this study is to demonstrate noninferiority in the visual acuity at distance when wearing Alcon serafilcon A contact lenses compared to ACUVUE® OASYS with HYDRACLEAR® PLUS Technology

| contact lenses when worn on a daily wear modality. |
|----------------------------------------------------|

At the end of the study, a clinical study report will be prepared in accordance with applicable regulatory requirements and standards.

#### 5.3 Risks and Benefits

The clinical investigation process risks are managed through appropriate training and monitoring according to the protocol specific monitoring plan. Investigational device risks, including risks associated with use of device and methods and procedures for application of device, are defined in the investigator's brochure and/or product labeling and are managed through review of safety assessments outlined in this protocol.

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of the test contact lens are features consistent with successful contact lens wear.

The Alcon serafilcon A contact lenses and AOHP contact lenses can be worn on daily wear modality until the end of their respective wear cycles.

A summary of the known potential risks and benefits associated with the investigational Alcon serafilcon A contact lens can be found in the investigator's brochure (see Package Insert for AOHP contact lenses). Risks are minimized by compliance with the eligibility criteria and study procedures, and through close supervision by a licensed clinician during exposure to the study lenses. The potential harms associated with on-eye exposure to the new lens materials include toxicity response, blurred vision, and ocular discomfort. In general, the risks with the investigational contact lens are anticipated to be similar to other marketed soft contact lenses.

The site personnel will educate subjects on proper hygiene and lens handling, and compliance with the use of contact lenses according to the protocol. Subjects should be instructed not to wear contact lenses while sleeping or swimming. The site personnel will also advise the subjects to remove contact lenses and return for prompt follow-up of symptoms, such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.

There may also be unknown risks to use of test product. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, clinical oversight, and monitoring

Refer to the IB for additional information.

#### 6 STUDY OBJECTIVES

#### 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

# The primary objective of this study is to demonstrate noninferiority in the visual acuity at distance when wearing Alcon serafilcon A contact lenses compared to AOHP contact lenses when worn in a daily wear modality. Endpoint(s) • Distance visual acuity (logMAR) with study lenses at Week 1

#### 6.2 Secondary Objective(s)

Not Applicable.





#### 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Describe the safety profile of the study products. | <ul><li>Adverse events</li><li>Biomicroscopy findings</li></ul> |
| | <ul> <li>Device deficiencies</li> </ul> |

#### 7 INVESTIGATIONAL PLAN

#### 7.1 Study Design

This will be a multisite, prospective, randomized, double masked, bilateral, crossover study comparing 2 reusable soft contact lenses. The expected duration of subject participation in the study is approximately 28 days (~14 days per each lens type), with 7 scheduled visits. Subjects will be asked to wear their habitual spectacles only (no contact lens wear) during the washout periods for 2 (at least 48 hours) to 4 days after Visit 1 and after Visit 4.



#### 7.2 Rationale for Study Design

This study design is justified based upon an evaluation of the results of relevant preclinical and clinical testing, as described within the IB.
The investigational contact lens is intended for the optical correction of refractive ametropia in persons with nondiseased eyes.

| The purpose of this study is to assess the clinical performance of the investigational Alcon serafilcon A contact lenses as compared to marketed AOHP contact lenses. |
|---|
| Procedures for measurement were selected based on common practice for these assessments. The design of this study is justified based upon preclinical and clinical testing, as described within the investigator's brochure. AOHP contact |
| lenses were chosen as the comparator product because these lenses also are reusable contact lenses (see Package Insert for AOHP contact lenses). |
| The intended use of this contact lens is vision correction; therefore, the measurement of distance VA is planned as the primary effectiveness endpoint. |
| The crossover design will ensure that the same subject is exposed to both the test and comparator lens materials; |
| The study will only include normal contact lens wearers to ensure the subjects participating in this trial represent the average clinic population and a population that can detect differences between lens materials. The study will exclude any current/habitual AOHP lens and daily disposable contact lens wearers, and any previous wearers of AOHP lens in the past 6 months prior to consent and any previous daily disposable contact lens wearers in the past 3 month prior to consent in order to reduce potential bias of wearers to their habitual contact lenses. |

# 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations

Status: Approved, Version: 3.0

Approved Date: 13 Apr 2023

Interim analysis will not be performed.

| 7.3 Rationale for Duration of Treatment/Follow | 7-U | p |
|------------------------------------------------|-----|---|
|------------------------------------------------|-----|---|

| Subjects will wear each study product bilaterally for their respective wear cycles on a daily |
|---|
| wear modality. |
| . The lenses will be provided by a qualified |
| unmasked study staff member in such a manner that the subject and the investigator remain |
| masked to the lens type. |

## 7.4 Rationale for Choice of Comparator Product

AOHP contact lenses were chosen as the comparator product because these lenses also are reusable contact lenses (see Package Insert for AOHP contact lenses).

## 7.5 Data Monitoring Committee

Not applicable.

#### **8 STUDY POPULATION**

Volunteer subjects aged 18 or over who are habitual spherical soft contact lens wearers (excluding current/previous ACUVUE® OASYS with HYDRACLEAR® PLUS Technology habitual lens wearers and daily disposable lens wearers), have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 8 hours per day.

One specific group of subjects will be recruited for this study: normal contact lens wearers.

The study population includes approximately 185 volunteer subjects to be enrolled at approximately ~14 sites, with approximately 14 subjects enrolled per site. The study population will consist of subjects with normal eyes (other than the need for optical correction for myopia), who are adapted, existing wearers of soft contact lenses in both eyes for at least the past 3 months and who wear contact lenses at least 5 days per week and at least 8 hours per day.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

- 1. Subject must be at least 18 years of age.
- 2. Subject must be able to understand and must sign an informed consent form (ICF) that has been approved by an Institutional Review Board (IRB).
- 3. Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
- 4. Manifest cylinder of  $\leq$  -0.75 D in each eye.
- 5. Best corrected visual acuity (BCVA) 20/25 Snellen (0.10 logMAR) or better in each eye.
- 6. Subject must possess spectacles and be willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.
- 7. Subject must be willing to stop wearing their habitual contact lenses for the duration of study participation.
- 8. Able to wear contact lenses within a range of sphere power from -1.00 D to -6.00 D (0.25 D steps) and subject willing and able to wear the study lenses for the full duration of the study.
- 9. Subject must be willing to wear contact lenses for at least 16 hours per day on the day prior to week 1 and on the day prior to week 2 follow up visits for both test and comparator lenses.

Status: Approved, Version: 3.0  Approved Date: 13 Apr 2023

10. Subject must be able to be successfully fit with test and comparator lenses.

#### 8.2 **Exclusion Criteria**

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

- 1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.
- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.
- 3. History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye.
- 4. Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study.
- 5. Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates.
- 6. Current or history of pathologically dry eye in either eye that, in the opinion of the investigator, would preclude contact lens wear.
- 7. Current or history of herpetic keratitis in either eye.
- 8. Eye injury in either eye within twelve weeks immediately prior to enrollment for this trial.
- 9. Current or history of intolerance, hypersensitivity, or allergy to any component of the study products.
- 10. Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.

- 11. Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear.
- 12. The investigator, his/her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of the aforementioned persons may not participate in the study.
- 13. Participation of the subject in a clinical trial within the previous 30 days or currently enrolled in any clinical trial.
- 14. Habitual AOHP contact lens wearers and current habitual wearers of any daily disposable contact lenses.

16. Currently pregnant, as stated by the subject

## 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

#### 9 TREATMENTS ADMINISTERED

## 9.1 Investigational Product(s)

Test Product(s): Alcon serafilcon A contact lenses

Comparator Product(s) (If ACUVUE® OASYS with HYDRACLEAR® PLUS

applicable): Technology contact lenses

#### Table 9–1 Test Product

| Test Product | Alcon serafilcon A contact lenses |
|---|---|
| Manufacturer | Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, Texas 76134-2099 USA |
| Indication for use and intended | The investigational contact lens is intended for the optical correction of refractive ametropia in persons with nondiseased eyes. |

| purpose in the | |
|---------------------|-----------------------------------------------|
| current study | |
| Product description | Material - serafilcon A |
| and parameters | • Water content $55 \pm 2\%$ |
| available for this | • Power range: -1.00 to -6.00 D in 0.25 steps |
| study | • Base curve (mm): 8.4 mm |
| | • Diameter (mm): 14.2 mm |

| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> </ul> </li> <li>Replacement lenses will not be provided to the subject. In the event a lens needs to be replaced, the subject must return to the site for a replacement lens. Until the replacement lens is obtained, the subject must store both study lenses in the provided lens care solution and wear their habitual spectacles.</li> <li>Exposure: Study lenses are to be worn during typical contact lens wearing hours, on all days during the study lens wearing period, at least 10 hours per day, over each treatment period (7 days (-0/+1) according to randomization assignment). Subjects will be asked to wear their study lenses for 16 hours on the days prior to each Follow-up Visit (Visit 3, 4, 6, &amp; 7).</li> <li>Lens Care: Cleaned and disinfected with CLEAR CARE®</li> </ul> |
|---|---|
| | Cleaning & Disinfecting Solution after each use. |
| Number/Amount of | Provided in bags of (25) lenses per power per bag |
| product to be | |
| provided to the site | |
| Packaging description | Blister foil pack |

| Labeling description | • Lens Foil label includes: |
|----------------------|----------------------------------------------------|
| | - material name and identifier |
| | - base curve |
| | - diameter |
| | - manufacturing protocol number |
| | <ul> <li>packing solution</li> </ul> |
| | - power |
| | - lot number |
| | - expiration date |
| | - content statement |
| | - investigational device statement |
| | - sponsor information |
| Storage conditions | Store at room temperature. |
| Lens Care | Cleaned and disinfected with CLEARCARE® Cleaning & |
| | Disinfecting Solution after each use. |
| Supply | Refer to the MOP for a detailed description |

Table 9–2 Comparator Product

| Comparator | ACUVUE® OASYS with HYDRACLEAR® PLUS Technology |
|---|---|
| Product(s) | contact lenses |
| Manufacturer | Johnson & Johnson Vision |
| Indication for Use | The comparator contact lens is intended for the optical correction of |
| | refractive ametropia in persons with nondiseased eyes |
| Product description | Material: senofilcon A |
| and parameters | • Water content: 38% |
| available for this | • Power range: -1.00 to -6.00 D in 0.25 steps |
| study | Base curve (mm): 8.4 mm and 8.8 mm |
| | • Diameter (mm): 14.0 mm |
| Formulation | See package insert for AOHP contact lenses |
| Usage | • Wear: |

| Number/Amount of Product to be Provided to the subject | <ul> <li>Daily Wear</li> <li>Bilateral</li> <li>Replacement lenses will not be provided to the subject. In the event a lens needs to be replaced, the subject must return to the site for a replacement lens. Until the replacement lens is obtained, the subject must store both study lenses in the provided lens care solution and wear their habitual spectacles.</li> <li>Exposure: Study lenses are to be worn during typical contact lens wearing hours, on all days during the study lens wearing period, at least 16 hours a week, over each treatment period (14 day (-0/+1) according to randomization assignment). Subjects will be asked to wear their study lenses for 16 hours a week prior to each Follow-up Visit (Visit 3, 4, 6, &amp; 7).</li> <li>Lens Care: Cleaned and disinfected with CLEAR CARE® Cleaning &amp; Disinfecting Solution after each use.</li> <li>Each Site will procure their own comparator lenses.</li> </ul> |
|---|---|
| Packaging description | Provided in commercial packaging |
| Labeling description | Commercial foil. |
| Storage conditions | Store at room temperature |
| Lens Care | Cleaned and disinfected with CLEAR CARE® Cleaning & Disinfecting Solution after each use. |
| Supply | <ul> <li>Refer to the MOP for a detailed description</li> <li>Each site will procure their own comparator lenses.</li> <li>CLEAR CARE® contact lens solution supplied by sponsor to be provided to the subject</li> </ul> |

# 9.2 Other Medical Device or Medication Specified for Use During the Study

During the clinical study, additional medical devices and/or medications that are required in conjunction with the treatment include the following:

- CLEAR CARE® Cleaning & Disinfecting Solution supplied by sponsor to be provided to subjects for use during the study.
- Lubrication/rewetting drops will not be permitted.

## 9.3 Treatment Assignment / Randomization

Subjects will be randomized in a 1:1 manner to receive treatment (lens) in crossover sequence: test product then comparator product or comparator product then test product, respectively.

| Sequence | EDC/randomization integration system | Lens Name |
|------------|--------------------------------------|-------------------------|
| Sequence 1 | LID022821/AOHP | Alcon serafilcon A/AOHP |
| Sequence 2 | AOHP/LID022821 | AOHP/Alcon serafilcon A |

Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

A randomization list will be generated using a validated system that automates the random assignment of treatment (lens sequence) to randomization numbers in the specified ratio. Subjects will be assigned treatment (lens sequence) according to the randomization list uploaded in the randomization system. The randomization list will be generated and maintained by the study sponsor

At Visit 1 after completion of BCVA (OD, OS, logMAR distance with manifest refraction), biomicroscopy, and fitting of investigational products (trial assessments for test and comparator) all eligible subjects will be randomized via the EDC/randomization integration system to one of the treatments (lens sequences). The investigator or delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject randomization list but will not be communicated to the site user. The EDC/randomization integration system will inform the site user of the treatment (lens sequence) assignment to be dispensed to the subject.

## 9.4 Treatment masking

This study is double masked with subjects randomized to use Alcon serafilcon A and AOHP for the duration of the two 2-week treatment periods.





In the event of a medical emergency where the knowledge of subject treatment is required, an individual investigator will have the ability to unmask the treatment assignment for a specific subject after contacting an appropriate study sponsor representative if time allows.

## 9.5 Accountability Procedures

Upon receipt of the IPs, the investigator or delegate must conduct an inventory. During the study, designated unmasked study staff must provide the IPs to the subjects in accordance with their randomization assignment. Throughout the study, the investigator or delegate must maintain records of IP dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the investigator must be accounted for by study sponsor personnel, and in no case be used in an unauthorized situation.

The investigator should make every effort to collect unused lenses, foils, and supplies from subjects.

It is the investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All unused products are available for return to the study sponsor, as directed

• Any study lenses or solutions associated with a device deficiency or with any product-related adverse event (i.e., ADE or SADE) are returned to the study sponsor for investigation, unless otherwise directed by the sponsor. Refer to Section 11 of this protocol for additional information on the reporting of device deficiencies and AEs and the return of study products associated with these events.

The investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.

#### 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications,
- Any medical procedure or hospitalization that occurred or is planned
- Any nondrug therapies (including physical therapy and blood transfusions).

The investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 7 office visits, as shown below.

| Visit # | Visit Type | Visit Window |
|---------|--------------------------|---------------------------------|
| Visit 1 | Screening/Baseline | N/A |
| Visit 2 | Dispense Lens 1 | 2 (at least 48 hours) - 4 |
| | | days after Visit 1 (Washout |
| | | period with habitual spectacles |
| | | only after Visit 1) |
| Visit 3 | Week 1 Follow-up Lens 1 | 7 -0/+ 1 days after Visit 2 |
| Visit 4 | Week 2 Follow- up Lens 1 | 7 -0/+ 1 days after Visit 3 |

| Visit 5 | Dispense Lens 2 | 2 (at least 48 hours) - 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4) |
|---|---|---|
| Visit 6 | Week 1 Follow-up Lens 2 | 7 -0/+ 1 days after Visit 5 |
| Visit 7 | Week 2 Follow-up Lens 2/Exit | 7 -0/+ 1 days after Visit 6 |

Unscheduled Visits and Early Exit Visits are allowed, if necessary.

Study lenses will be provided to the subjects to take home for daily wear during the course of the trial.

Study randomization will occur at Visit 1 to determine assigned lens sequence. Subjects will be provided the assigned lenses to take home at Visit 2, Visit 3, Visit 5 and Visit 6. Study contact lens fitting will occur at Visit 1 for both study lenses. If a subject cannot be successfully fit (either study lens) according to the study lens fitting guides as determined by the investigator, they will be required to exit from the study.

Lubrication/rewetting drops will not be permitted during this study.

#### 10.1 Informed Consent and Screening

The investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF before any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.

The investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

#### **10.2 Description of Study Procedures and Assessments**

Study-specific procedures and assessments described here may include standard of care; other standard of care procedures performed in the clinical management of the subject are not excluded.

Detailed descriptions of assessments and procedures are provided in the MOP. The investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

#### 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

## **10.2.2** Medical History

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

Medical History and Concomitant Medications will be collected in the eCRF as outlined in the MOP

## 10.2.3 Investigational Product Compliance

Review subject compliance with the IP usage and adjunct product usage and collect all used and unused study IPs and other products that were dispensed.

## 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any adverse events that are observed or reported since the previous visit, including those associated with changes in concomitant medication dosing in the subject source documents. See Section 11 for further details regarding AE collection and reporting.

## 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment

SLE of the cornea, iris/anterior chamber and lens must be performed in both eyes before instillation of any diagnostic eye drops.

#### 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11.

#### 10.2.7 Best Corrected Visual Acuity: Safety Assessment

LogMAR visual acuity testing for both eyes must be performed prior to any assessment requiring administration of eye drops to dilate the eyes, or any assessment requiring contact with the eye.

#### 10.3 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visit and the visit is conducted by study personnel, this visit must be documented as an unscheduled visit. If the subject seeks medical attention outside the clinic (for example, at an emergency room) or at the clinic but is seen by non-study personnel, the investigator is to capture adverse event-related information on the Adverse Event form upon becoming aware.

During all unscheduled visits, the investigator must conduct the following procedures:

- Collect adverse event information
- Collect Device Deficiency information
- Record changes in medical condition or concomitant medication
- Biomicroscopy
- Review lens wear calendar

The investigator may perform additional procedures for proper diagnosis and treatment of the subject. The investigator must document this information in the subject's case history source documents.

If during an unscheduled visit the subject is discontinuing the IP or discontinuing from the study, the investigator must conduct Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments and Section 10.4.3, as possible.

#### 10.4 Discontinued Subjects

#### 10.4.1 Screen Failures

Subjects who were excluded from the study after signing the informed consent and prior to randomization to IP.

The investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be reused.

#### 10.4.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the investigator after signing the informed consent, including screen failures.

Subject numbers of discontinued subjects must not be reused (i.e., subject replacement is not allowed).

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the investigator, continued treatment poses a risk to their health.

For subjects discontinuing from the study, the investigator must complete all Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments and Section 10.4.3, if the subject is willing and able, and if in the opinion of the investigator it is safe for the subject to do so.

The investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an Early Exit Visit. Refer to Table 3-1 and the MOP for details.

#### 10.5 Clinical Study Termination

The study sponsor reserves the right to suspend or close the investigational site or suspend or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the study sponsor:

- The study sponsor must:
  - Immediately notify the investigator(s) and subsequently provide instructions for study termination.
  - Inform the investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for poststudy treatment options as needed.

The investigator may terminate the site's participation in the study for reasonable cause.

Breaking of the masked treatment codes will be done after locking the database.

## 10.5.1 Follow-Up of Subjects After Study Participation has Ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (Test Product).

Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11-1 Categorization of All Adverse Events



Status: Approved, Version: 3.0

Approved Date: 13 Apr 2023

Figure 11-2 Categorization of All Serious Adverse Events



#### **Specific Events Relevant to this Protocol**

#### Serious Adverse Events

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics:
  - Central or paracentral location
  - o Penetration of Bowman's membrane

- Infiltrates >2 mm diameter
- o Iritis
- Increase in intraocular pressure
- Culture positive for microorganisms
- Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon
- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

#### Significant Non-Serious Adverse Events

A significant non-serious AE is a device-related, non-sight threatening adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. In addition, the investigator must report any occurrence of the following as a Significant Non-Serious Adverse Event:

- Peripheral non-progressive non-infectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score greater than or equal to grade 3 (Refer to MOP for grading scales) [Grading scale is based on ISO 11980:2012 unless specified differently in MOP]
- Temporary vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that persists for 2 or more weeks
- Neovascularization score greater than or equal to grade 2 (Refer to MOP for grading scales) [Grading scale is based on ISO 11980:2012 unless specified differently in MOP]

The above events are based on the categories provided in the ISO 11980 and the US FDA Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses and Contact Lens Care Products.

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with patient harm (i.e., ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any patient harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (e.g., incorrect lens power/diameter/base curve/color)
- Lens/solution cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (e.g., mislabeled product, tampered seal, leaking bottle/container)
- Suspect product contamination

## 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the investigator should inquire about AEs by asking the standard questions shown below and report as applicable:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take because of a new health issue since your last study visit?"

In addition, changes in *any protocol-specific parameters* evaluated during the study are to be reviewed by the Investigator. Any untoward (unfavorable and unintended) change in *a protocol-specific parameter or questionnaire response* that is clinically relevant, in the opinion of the Investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

#### 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any preexisting medical conditions or signs/symptoms present in a subject prior to the start of the study (i.e., before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

For each recorded event, the ADEs and SAEs documentation must include date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. Furthermore, the investigator must document all device deficiencies reported or observed with test and control products on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the study sponsor immediately as follows:

- ADEs or SAEs are documented on the *Serious Adverse Event and Adverse Device Effect* eCRF within 24 hours of the investigator's or site's awareness.
- Device deficiencies are documented on the *Device Deficiency* eCRF within 24 hours of the investigator's or site's awareness.
- A printed copy of the completed *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate source form.
- Document all relevant information from Discharge Summary, Autopsy Report,
- Certificate of Death etc., if applicable, in narrative section of the *Serious Adverse Event and Adverse Device Effect* eCRF.

Note: Should the EDC system become non-operational, the site must complete the appropriate paper Serious Adverse Event and Adverse Device Effect and/or Device Deficiency Form. The completed form is emailed to the Study Sponsor at msus.safety@Alcon.com according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

In addition to recording all AEs into the EDC system, any AEs and device deficiencies for non-study marketed devices/products (e.g., CLEAR CARE® Cleaning & Disinfecting Solution used concomitantly during the study will be considered and processed as spontaneous following the postmarket vigilance procedures) and should be communicated to the device's/product's manufacturer as per local requirements.

Study sponsor representatives may be contacted for any protocol related question and their contact information is provided in the Manual of Procedures that accompanies this protocol.

*Note:* depending upon the nature of the AE or device deficiency being reported, the study sponsor may request copies of applicable portions of the subject's medical records. The investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

#### **Intensity and Causality Assessments**

Where appropriate, the investigator must assess the intensity (severity) of the AE based on medical judgment with consideration of any subjective symptom(s), as defined below:

#### **Intensity (Severity)**

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the subject's inability to work or engage in their usual activities.

For every AE in the study, the investigator must assess the causality (related or not related to the medical device or study procedure). An assessment of causality will also be performed by study sponsor utilizing the same definitions, as shown below:

#### **Causality**

Related An AE classified as related may be either definitely related or possibly related where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply unlikely to be related (i.e., there are other more likely causes for the AE).

The study sponsor will assess the AEs and may upgrade the investigator's assessment of seriousness and/or causality. The study sponsor will notify the investigator of any AEs that is upgraded from non-serious to serious or from unrelated to related.

#### 11.4 Return Product Analysis

Study sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.

Alcon study products associated with device deficiencies and/or product related AEs should be returned and must include the Complaint # which will be provided by study sponsor after the case is entered in the study sponsor's Global Product Complaint Management System (GPCMS).

### 11.5 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study Reference Section 9.4 for details on masked and unmasked persons. If the treatment code needs to be broken in the interest of subject safety, the investigator is encouraged to contact an appropriate study sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (i.e., medical emergency), the code may be broken prior to contact with the study sponsor. The study sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the study sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements.

## 11.6 Follow-Up of Subjects with Adverse Events

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The investigator should provide the study sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of discontinuation, any additional information received at follow-up should be documented in the eCRFs up to study completion (i.e., database lock). Any additional data received up to 3 months after subject completed the study should be documented and available upon the study sponsor's request.

All complaints received after this time period will be considered and processed as spontaneous (following the post-market vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements. The investigator should also report complaints on non-Alcon products directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

## 11.7 Pregnancy in the Clinical Study

Women who are pregnant (as stated by the subject) at the time of study entry are excluded from participation. However, pregnancy should be included in the corresponding eCRF if a woman becomes pregnant (as stated by the subject) during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case—by-case basis.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum, as well as confidence intervals (CIs) or confidence limits where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

## 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens sequence) assignment and locking the database, based upon the Deviations and Evaluability Plan (DEP).

## 12.2 Analysis Sets

## 12.2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study,

For treatment-

emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

#### 12.2.2 Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses

evaluated in this study.

### 12.2.3 Per Protocol Analysis Set

The per protocol (PP) analysis set is a subset of FAS and excludes all data/subjects that have met any of the critical deviation or evaluability criteria identified in the DEP.

#### 12.3 Demographic and Baseline Characteristics

Demographic information will be summarized by lens sequence and overall. Frequencies and percentages will be presented for categorical variables such as sex, age group, race, and ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.



## 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to demonstrate noninferiority in the VA at distance when wearing Alcon serafilcon A contact lenses compared to AOHP contact lenses when worn on a daily wear modality.

The primary endpoint is distance VA with study lenses at Week 1, collected for each eye in logMAR.

#### **12.4.1.1** Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

$$H_0$$
:  $\mu_{(T)} - \mu_{(C)} \ge 0.05$   
 $H_a$ :  $\mu_{(T)} - \mu_{(C)} < 0.05$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA at Week 1 for Alcon serafilcon A and AOHP, respectively, on the logMAR scale.

### 12.4.1.2 Analysis Methods

A mixed effects repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, period, sequence, visit, and lens by visit interaction. Within subject correlation due to eye and crossover will also be accounted for in the model. Lens difference (Alcon serafilcon A minus AOHP) and the corresponding one-sided 95% upper confidence limit (UCL) will be computed at Week 1. Noninferiority will be declared if the UCL is less than 0.05.







#### 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for

#### 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device Deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (frequencies and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (last assessment prior to study lens exposure) to any subsequent visit within the same period will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits within the same period for those eyes experiencing the increase.

Two listings for device deficiencies, prior to exposure to study contact lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be conducted for the safety analyses.

## 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

## 12.8 Sample Size Justification

Sample size calculation is based on a prior clinical study (which evaluated performance of Alcon serafilcon A and AOHP.







### 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

## 13.1 Subject Confidentiality

The investigator must ensure that the subject's identity is kept confidential throughout the course of the study. In particular, the investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. The study sponsor may collect a copy of the enrollment log without any directly identifying subject information.

## 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the study sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility

- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The principal investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number, and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

## 13.4 Sponsor and Monitoring Responsibilities

The study sponsor will select principal investigators that are qualified by education, training, and experience to assume responsibility for the proper conduct of this clinical trial.

The study sponsor is financially funding this clinical trial and will compensate the investigator and/or the institution(s) at which the study is conducted in accordance with a signed clinical trial agreement.

The study sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate study sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written and fax correspondence. Close out visits will take place after the last visit of the last subject at the site.

A coordinating investigator may be identified by the study sponsor to review and endorse the final study report. In cases where a coordinating investigator is engaged, the study sponsor will select the coordinating investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

#### 13.5 Regulatory Documentation and Records Retention

The investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the study sponsor and the investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.

Additionally, the investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the study sponsor. If the investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the study sponsor must be notified, and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

## 13.6 Quality Assurance and Quality Control

The study sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the study sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the study sponsor

with the investigator/institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

Investigations are conducted in compliance with Good Clinical Practices; international and national regulations, laws and guidelines; the conditions of approval imposed by reviewing IRBs/IECs or regulatory authorities; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki and Good Clinical Practices outlined within ISO 14155.

- The SOPs of the study sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations shall apply.
- Notifications and timelines for reporting protocol deviations should be based upon applicable Ethics Committee requirements.

The investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. The investigator is not allowed to deviate from the protocol except to protect the rights, safety, and well-being of human subjects under emergency circumstances. Emergency deviations may proceed without prior approval of the sponsor and the IRB/IEC but shall be documented and reported to the sponsor and the IRB/IEC as soon as possible. Deviations from this protocol, regulatory requirements, and/or GCP must be recorded and reported to the sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Failure to implement identified corrective and preventative actions may result in site closure by the sponsor. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC. The investigator must provide documentation of the IRB/IEC approval to the study sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the Package Insert, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. Any additional requirements imposed by the IEC or regulatory authority shall be followed. At the end of the study, the investigator must notify the IRB/IEC about the study's completion. The IRB/IEC

also must be notified if the study is terminated prematurely. Finally, the investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject. The obtaining of consent shall be documented before any procedure specific to the clinical investigation is applied to the subject.

The investigator must have a defined process for obtaining the required consent. Specifically, the investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the investigator, and if required by local regulation, other qualified personnel. The investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and sponsor-designated personnel. The investigator must keep the original, signed copy of the consent (file in subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

The study sponsor assures that the key designs of this protocol will be registered on public databases where required by current regulations, and, as applicable, results will be posted.

#### **15 REFERENCES**

## 15.1 Regulations and Standards

The following references may be applicable in whole or in part for this clinical trial.

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- EN ISO 14155:2020 Clinical Investigation of Medical Devices for Human Subjects -Good Clinical Practice
- 21 CFR Part 11 Electronic Records; Electronic Signatures

- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators





